CLINICAL TRIAL: NCT02960815
Title: Safety and Immunogenicity of Seasonal Influenza Vaccine With Topical Imiquimod in Immunocompromised Patients: A Randomized Controlled Pilot Trial
Brief Title: Imiquimod and Influenza Vaccine for Immunocompromised Patients
Acronym: IMIFLU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Oriol Manuel, PD Dr, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-01540
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Influenza Vaccine
Keywords: influenza vaccine; Transplantation; imiquimod; HIV infection; immunogenicity
MeSH Terms: conditions — Influenza, Human; HIV Infections | interventions — mutagrip; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intramuscular vaccine (Active Comparator): The control intervention consists in the administration of the standard intramuscular influenza vaccine (Mutagrip®), containing 15 μg of each of the three viral strains without imiquimod.
  Interventions: Biological: Mutagrip
- Imiquimod and intradermal vaccine (Experimental): In the imiquimod and intradermal vaccine arm, intervention consists in the topical application of a single bag of Aldara™ creme 5%, containing 12.5 mg of imiquimod, on a 16 cm2 square delimitated area on the non-dominant arm at the time of influenza vaccination. An intradermal influenza vaccine preparations containing 15 μg of each of the three viral strains (Intanza®) will be administrated in the centre of the marked area after the imiquimod cream is fully absorbed.
  Interventions: Biological: Intanza; Drug: Aldara
- Imiquimod and intramuscular vaccine (Experimental): In the imiquimod and intramuscular vaccine arm, intervention consists in the topical application of a single bag of Aldara™ creme 5%, containing 12.5 mg of imiquimod, on a 16 cm2 square delimitated area on the non-dominant arm at the time of influenza vaccination. An intramuscular influenza vaccine preparations containing 15 μg of each of the three viral strains (Mutagrip®) will be administrated in the centre of the marked area after the imiquimod cream is fully absorbed.
  Interventions: Biological: Mutagrip; Drug: Aldara

INTERVENTIONS:
Biological: Intanza
  Arms: Imiquimod and intradermal vaccine
Biological: Mutagrip
  Arms: Imiquimod and intramuscular vaccine; Intramuscular vaccine
Drug: Aldara
  Arms: Imiquimod and intradermal vaccine; Imiquimod and intramuscular vaccine

SUMMARY:
In this open label, single centre, pilot randomized controlled clinical trial the investigators aim to compare the immunogenicity and safety of a new influenza vaccination strategy consisting in the topical administration of imiquimod at the injection site before vaccination vs. a standard intramuscular vaccine injection in SOT recipients and HIV-infected individuals. The investigators planned to enroll 70 outpatients patients (50% solid-organ transplant recipients and 50% HIV-infected patients) regularly followed at the Transplantation center and the Infectious disease outpatients' clinics of the Lausanne University Hospital. Study participants will be randomized in a 1:1:1 ratio to receive the standard intramuscular vaccine (control group) or a topical application of an imiquimod containing cream followed by intramuscular (imiquimod-IM) or intradermal (imiquimod-ID) vaccine injection. After vaccination participants will be followed for a period of 180 days. Blood samples will be drawn at baseline and at day 21 and 180 for assessment of immunogenicity. Safety outcomes will be assessed immediately after vaccine administration, and at day 7 (phone call), 21 and 180.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written, informed consent
* Age > 18 years
* HIV infection or at least 3 months after kidney transplantation
* Stable outpatients
* Able and willing to comply with the study protocol

Exclusion Criteria:

* Documented egg and/or imiquimod allergy
* Previous life-threatening reaction to seasonal influenza vaccine (i.e. Guillain-Barré Syndrome)
* Previous severe reaction to imiquimod cream
* Pregnancy or breast-feeding
* Patients with autoimmune diseases
* For HIV-infected patients:

  * Current active opportunistic infection
* For kidney transplant recipients:

  * Ongoing therapy for rejection (including steroid pulse or prednisone > 2 mg/kg/day over more than 14 days)
  * Ongoing therapy with IVIG and eculizumab or current and past (<6months) therapy with rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Response to the vaccine | 21 days after vaccination
  Vaccine response rate (=seroconversion rate) at day 21 is the proportion of participants exhibiting a fourfold or greater increase of anti haemagglutinin (anti-HA) antibodies from baseline, measured by haemagglutinin inhibition (HI) assay 21 days after vaccination, for at least one viral strain.

SECONDARY OUTCOMES:
Seroprotection rates | Baseline, 21 and 180 days after vaccination
  Seroprotection rates for each vaccine strain at baseline, and 21 and 180 days after vaccination. Seroprotection rate is defined as the proportion of patients exhibiting an anti-HA antibody titer of 1:32 or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Manuel, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manuel O, Pascual M, Hoschler K, Giulieri S, Alves D, Ellefsen K, Bart PA, Venetz JP, Calandra T, Cavassini M. Humoral response to the influenza A H1N1/09 monovalent AS03-adjuvanted vaccine in immunocompromised patients. Clin Infect Dis. 2011 Jan 15;52(2):248-56. doi: 10.1093/cid/ciq104. PMID 21288852
- [Result] Cordero E, Manuel O. Influenza vaccination in solid-organ transplant recipients. Curr Opin Organ Transplant. 2012 Dec;17(6):601-8. doi: 10.1097/MOT.0b013e3283592622. PMID 23042206
- [Result] Manuel O, Humar A, Berutto C, Ely L, Giulieri S, Lien D, Meylan PR, Weinkauf J, Pascual M, Nador R, Aubert JD, Kumar D. Low-dose intradermal versus intramuscular trivalent inactivated seasonal influenza vaccine in lung transplant recipients. J Heart Lung Transplant. 2011 Jun;30(6):679-84. doi: 10.1016/j.healun.2011.01.705. Epub 2011 Mar 5. PMID 21377898